CLINICAL TRIAL: NCT00218881
Title: An Effective Alternative to the Standard Referral System for HIV Testing in the ED
Brief Title: An Effective Alternative to the Standard Referral System for HIV Testing in the Emergency Department During Off Hour Tours: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Bronx Healthcare Network (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 03-090
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2005-10-25 (Estimated); Status verified 2005-09

CONDITIONS: HIV Counseling and Testing; HIV Infections
Keywords: HIV prevention; HIV screening; Emergency Medicine; HIV counseling and Testing; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Procedure: HIV educational video

SUMMARY:
To compare HIV testing rates in ED patients offered video-assisted informed consent off-hours versus those referred to an HIV counselor the next business day.

DETAILED DESCRIPTION:
ED-based HIV counseling and testing (C&T) is in its early stages of development. Most urban ED patients requesting or requiring HIV testing are referred to C&T sites that are usually available only during regular business hours. Patient compliance with these referrals has been disappointing.

To improve ED access to HIV testing, we developed a video alternative to in-person pre-test counseling to provide the fundamental elements of the counseling. The video was based on the educational elements required by the New York State Department of Health (DOH) for HIV pre-test counseling. In a previous study, we demonstrated that the educational video performed as well as live counselors in conveying the information needed for inner city ED patients to consent to HIV testing. The present study was designed to compare HIV testing rates in ED patients offered video-assisted informed consent for HIV testing versus the standard referral for live C&T the next business day.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years and older were approached while waiting for ED provider.

Exclusion Criteria:

* Patients who were clinically unstable
* Unable to understand the consent process
* Had been HIV tested within 6 months and were informed of the result, or had a confirmed diagnosis of HIV were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408
Dates: Start 2003-10; Study Completion 2004-07

PRIMARY OUTCOMES:
HIV testing rates in ED patients offered video-assisted informed consent off-hours versus those referred to an HIV counselor the next business day.

SECONDARY OUTCOMES:
Comparing return rates for HIV results in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD<MS, Principal Investigator — North Bronx Healthcare Network, Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States